CLINICAL TRIAL: NCT02693691
Title: CardioMEMS European Monitoring Study for Heart Failure
Acronym: MEMS-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10105
Record Dates: First submitted 2016-02-20; First posted 2016-02-29 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CardioMEMS HF System (Experimental): Subjects will collect pulmonary artery pressure measurements daily which will be used by health care professionals to adjust cardiac medications.
  Interventions: Device: CardioMEMS HF System

INTERVENTIONS:
Device: CardioMEMS HF System — Pulmonary Artery Pressure Monitoring

SUMMARY:
The purpose of this study is to characterize the use of the CardioMEMS™ HF System when used in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Indicated to receive a CardioMEMS sensor implant per the CardioMEMS™ HF System User's Manual
* ≥ 18 years of age
* Diagnosis of New York Heart Association (NYHA) Class III Heart Failure at the time of sensor implantation
* Hospitalization for worsening HF, as defined in the protocol, within 12 months prior to the CardioMEMS HF System implant
* Subjects with reduced Left Ventricular Ejection Fraction (LVEF) must be on stable Guideline Directed Medical Therapy (GDMT) as tolerated
* Written informed consent obtained from subject

Exclusion Criteria:

* Known coagulation disorders or inability to take two types of blood thinning medications for one month after the sensor is implanted
* Subjects deemed a candidate for transplant, Ventricular Assist Device, or hospice care in the next 12 months or are otherwise not expected to be able to complete the study follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03-31 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Angermann, Prof. Dr., Principal Investigator — Deutsches Zentrum für Herzinsuffizienz Würzburg; Michael Boehm, Prof. Dr., Principal Investigator — University Hospital, Saarland
Locations (2):
- Germany (2):
  - Klinukum Coburg, Coburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zile MR, Abraham WT, Stevenson LW, Costanzo MR, Angermann CE, Mehra MR, Desai AS, Ducharme A, Johnson N, Henderson J, Lindenfeld J. Relationship Between Remote, Ambulatory Pulmonary Artery Pressures, and All-Cause Mortality in Patients With Chronic Heart Failure. Circ Heart Fail. 2025 Jun;18(6):e012754. doi: 10.1161/CIRCHEARTFAILURE.124.012754. Epub 2025 Apr 14. PMID 40223608
- [Derived] Bohm M, Assmus B, Anker SD, Asselbergs FW, Brachmann J, Brett ME, Brugts JJ, Ertl G, Wang A, Hilker L, Koehler F, Rosenkranz S, Leistner DM, Abdin A, Wintrich J, Zhou Q, Adamson PB, Angermann CE. Less loop diuretic use in patients on sacubitril/valsartan undergoing remote pulmonary artery pressure monitoring. ESC Heart Fail. 2022 Feb;9(1):155-163. doi: 10.1002/ehf2.13665. Epub 2021 Nov 4. PMID 34738340
- [Derived] Angermann CE, Assmus B, Anker SD, Brachmann J, Ertl G, Kohler F, Rosenkranz S, Tschope C, Adamson PB, Bohm M. Safety and feasibility of pulmonary artery pressure-guided heart failure therapy: rationale and design of the prospective CardioMEMS Monitoring Study for Heart Failure (MEMS-HF). Clin Res Cardiol. 2018 Nov;107(11):991-1002. doi: 10.1007/s00392-018-1281-8. Epub 2018 May 19. PMID 29777373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 239 subjects at 31 investigational sites in Germany, The Netherlands, and Ireland. The first subject was enrolled on 13 May 2016 and the last subject was enrolled on 29 March 2018. The last 12-month follow-up was completed on 19 March 2019. Data was collected until the database closure date, 28 June 2019.
Pre-assignment Details: Three of the 239 subjects enrolled withdrew before implantation was attempted. Of the 236 subjects who had an attempted implant, two subjects were not implanted. One subject was not implanted because there was a failure to meet screening criteria and the other subject experienced an AE during the implant procedure and was not implanted.
Period: Primary Endpoint Analysis (First 12M)
Arm/Group | CardioMEMS HF System
Started | 234
Completed | 184
Not Completed | 50
Not completed — Death | 30
Not completed — Withdrawal by Subject | 12
Not completed — Physician Decision | 7
Not completed — Adverse Event | 1
Period: Extended Follow-Up (Until Last pt 12M)
Arm/Group | CardioMEMS HF System
Started | 184
Completed | 160
Not Completed | 24
Not completed — Death | 12
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | CardioMEMS HF System
Number analyzed (Participants) | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 186
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 216
  Netherlands | 19
  Ireland | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (5.3)
Ejection Fraction [Count of Participants; unit: Participants] — Ejection fraction (EF) is a measurement of the percentage of blood leaving the heart each time it contracts. Heart failure patients with an EF <40% are considered to have reduced ejection fraction (HFrEF) where as patients with an EF >=40% are considered to have preserved ejection fraction (HFpEF).
  Participants
    HFrEF (EF < 40%) | 168
    HFpEF (EF ≥ 40%) | 68
    Unknown | 3
HF Etiology [Count of Participants; unit: Participants]
  Ischemic Cardiomyopathy | 128
  Non-Ischemic Cardiomyopathy | 87
  Unknown | 24

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Device/System Related Complications
Description: This primary safety endpoints is freedom from device/system related complications (DSRCs) which is defined as an adverse event that is, or is possibly, related to the device/system (wireless pressure sensor or external electronics) and has at least one of the following characteristics: is treated with invasive means (other than intramuscular medication or right heart cauterization which is used for diagnostic purposes); results in death of the subject; or results in the explant of the device. The pre-specified goal of this endpoint was was to have a freedom from DSRC greater than 0.80 at 12 months post-implant.
Time Frame: one year
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CardioMEMS HF System
Number analyzed (Participants) | 239
percentage of patients | 98.3 [95.8 to 100]

2. Primary Outcome: Freedom From Pressure Sensor Failure
Description: This primary safety endpoints is freedom from pressure sensor failure greater than 0.90 at 12 months post-implant.
Time Frame: one year
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CardioMEMS HF System
Number analyzed (Participants) | 239
percentage of patients | 99.6 [97.6 to 100]

3. Primary Outcome: Percent of Successful Pulmonary Artery Pressure Data Transmissions
Description: Patient data transmission success is defined as the percentage of successful transmissions among attempted transmissions. All subjects who were consented and implanted with a pressure sensor regardless of study completion status are included in this analysis. All attempted data transmissions through the 12-month visit or death or withdrawal are included in the analysis. For each subject, the patient data transmission success rate (% of successful transmission) was calculated as total number of successful transmissions divided by total attempted transmissions within 12 months.
Time Frame: one year
Population: All subjects who were consented and implanted with a pressure sensor regardless of study completion status were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of successful transmissions
Arm/Group | CardioMEMS HF System
Number analyzed (Participants) | 234
percentage of successful transmissions | 91.7 (13.0)

4. Secondary Outcome: Heart Failure Hospitalization (HFH) Rate
Description: Comparison of the annualized heart failure hospitalization (HFH) rate (including recurrent events) at 12 months post-implant with the rate (including recurrent events) 12 months prior to implant.
Time Frame: one year
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | CardioMEMS HF System
Number analyzed (Participants) | 234
Hazard Ratio | 0.38 [0.31 to 0.48]

ADVERSE EVENTS:
Time Frame: AEs were collected starting from enrollment and until the last patient completed 12 months follow-up.
Description: Non-serious Adverse Events were not collected as part of the protocol.
Arm/Group | CardioMEMS HF System
All-Cause Mortality (participants affected / at risk) | 42/234
Serious Adverse Events (participants affected / at risk) | 184/239
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CardioMEMS HF System (N=239)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 6 (10)
Abnormal heart rate or rhythm (Cardiac disorders) | 43 (61)
Decompensated HF (Cardiac disorders) | 103 (190)
Other cardiac disorders (Cardiac disorders) | 57 (85)
Endocrine disorders (Endocrine disorders) | 9 (9)
Gastrointestinal disorders (Gastrointestinal disorders) | 21 (24)
General disorders (General disorders) | 38 (49)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2)
Immune system disorders (Immune system disorders) | 2 (2)
Infection (Infections and infestations) | 51 (72)
Other infections and infestations (Infections and infestations) | 8 (8)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 19 (22)
Investigations (Investigations) | 6 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Nervous system disorders (Nervous system disorders) | 5 (5)
Renal failure (Renal and urinary disorders) | 34 (43)
Other renal and urinary disorders (Renal and urinary disorders) | 4 (4)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1)
Vascular disorders (Vascular disorders) | 17 (21)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 9 (11)
Eye disorders (Eye disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02693691/Prot_SAP_ICF_000.pdf